CLINICAL TRIAL: NCT00714480
Title: Thymoglobulin: Presence and Affect in the Central Lymphatic Compartment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: William H Marks MD PhD, Swedish Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: TMG 617
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Renal Transplantation; Immunosuppression
Keywords: Thymoglobulin; Renal Transplant; Kidney Transplant; Immunosuppression; Induction therapy
MeSH Terms: interventions — Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Other): Administration of anti-thymocyte globulin post-operative days -6,-4,-2, and 0
  Interventions: Drug: anti-thymocyte globulin
- Group II (Other): Administration of anti-thymoglobulin post-operative days -2, 0, 2 and 4
  Interventions: Drug: anti-thymocyte globulin
- Group III (Other): Administration of anti-thymocyte globulin post-operative days 0, 2, 4 and 6
  Interventions: Drug: anti-thymocyte globulin

INTERVENTIONS:
Drug: anti-thymocyte globulin — Administration of anti-thymocyte globulin at post-operative days -6, -4, -2 and 0
  Other Names: Thymoglobulin
  Arms: Group I
Drug: anti-thymocyte globulin — anti-thymocyte globulin post-operative days -2, 0, 2 and 4
  Other Names: Thymoglobulin
  Arms: Group II
Drug: anti-thymocyte globulin — Post-operative days 0, 2, 4 and 6
  Other Names: Thymoglobulin
  Arms: Group III

SUMMARY:
This study proposes to examine the effect of TMG therapy upon the cellular elements within the central (bone marrow) and peripheral (lymph node) lymphoid compartments of humans. Briefly, bone marrow aspirates and lymph nodes will be obtained at the time of transplant, from renal transplant recipients receiving TMG induction therapy. For comparative purposes, peripheral blood samples will also be obtained. Lymphocytes from these compartments will be assessed for CD antigen expression, apoptosis, cytokine production following memory immune responses, and functional assays to assess potential regulatory T-cell (Treg) activity.

DETAILED DESCRIPTION:
Polyclonal anti-thymocyte globulins are used with increasing frequency to induce immunosuppression in organ transplant recipients. Induction therapy is used for the majority of persons receiving kidney transplant. In 2004, 72% of patients that received a kidney transplant also received induction therapy. This number is up from 46% reported in 1995. Anti-Thymocyte Globulin is the most commonly used agent for induction therapy. It was used for 37% of kidney recipients in 2004, and its use appears to be increasing year over year. A prominent example of this class of drugs is Thymoglobulin(TMG), a purified, pasteurized gamma immune globulin, which is obtained by immunization of rabbits with human thymocytes. The resulting preparation contains polyclonal antibodies directed against multiple T-cell markers, including CD antigens, HLA, and homing receptors.

Although the mechanism of action for the immunosuppressive effects of TMG has not been fully elucidated, there is evidence that complement-dependent cell lysis and depletion, cell-surface antigen modulation, blocking of adhesion molecules, and partial T-cell activation/anergy may play potential roles.

Many of the effects of TMG are evident in the peripheral blood compartment, including a rapid decline in circulating T-cells. Non-human primate studies have demonstrated that TMG treatment leads to depletion of T-cells via apoptosis in peripheral lymphoid tissues (spleen and lymph nodes), but no studies have been conducted to assess the effect of TMG in the bone marrow, and no studies have examined the peripheral lymphoid tissue in humans receiving TMG therapy.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects age 18 years or older who qualify to receive a living (related or unrelated) kidney allograft using steroid free induction immunosuppression.
2. Single organ recipient (kidney only)
3. Subjects receiving first renal transplant
4. Women of childbearing potential should have a negative serum pregnancy test within 1 week prior to beginning study medications
5. Subjects with no prior history of immunosuppression
6. Subjects with no systemic illness (i.e. diabetes, autoimmune disease)
7. Subjects with negative serologies (Hep B, Hep C, HIV)
8. Subjects who are candidates for TMG induction
9. Subjects providing written consent
10. Subjects who are compliant and able to complete all the assessment procedures

Exclusion Criteria:

1. Subjects less than 18 years of age
2. Subjects who do not meet criteria for steroid free protocol
3. Subjects who are pregnant, lactating or nursing
4. Child bearing women not willing to use a reliable form of contraception
5. Subjects with a known allergy to rabbits or rabbit products
6. Subjects receiving other medications considered to be experimental

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary objectives of this pilot study are to examine lymphocyte marker expression, quantitate specific lymphocyte subsets and apoptosis, and assess immune function in subjects receiving TMG. | Pretransplant days -6, -4, -2, 0; Post-transplant days 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: William H Marks, MD PhD, Principal Investigator — Swedish Medical Center; Paul Warner, PhD, Principal Investigator — Bloodworks
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States